CLINICAL TRIAL: NCT04107363
Title: The Effect of Oropharyngeal Aspiration Before Position Change on Reducing the Incidence of Ventilator-Related Pneumonia
Brief Title: Oropharyngeal Aspiration to Reduce Ventilator-Related Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe AKBIYIK (Other)
Responsible Party: Sponsor-Investigator, Ayşe AKBIYIK, Doctor of Philosophy (PhD) Research Assistant, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EGE.0.20.05.00/EY/739/924
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Ventilator-associated Bacterial Pneumonia
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: (Experimental): Patients in the experimental group underwent oropharyngeal aspiration prior to each position change in addition to routine nursing care (Endotracheal aspiration in case of indication and oropharyngeal aspiration in the follow-up; routine and non-routine position changes every 2 hours during the day and 4 hours during the night; oral care).
  Patients in this group underwent oropharyngeal aspiration at least 9 times in 24 hours with a pressure of 100-120 mmHg for 10 seconds prior to routine (2 hours a day, 4 hours a night) and non-routine position changes.
  After the oropharyngeal aspiration was completed, the patient's position was changed.
  Interventions: Procedure: Oropharyngeal aspiration before changing the position of the patient
- Control group (Other): The patients in the control group received routine nursing care in the unit. (Endotracheal aspiration in case of indication and oropharyngeal aspiration in the follow-up; routine and non-routine position changes every 2 hours during the day and 4 hours during the night; oral care).
  Interventions: Other: Control group:

INTERVENTIONS:
Procedure: Oropharyngeal aspiration before changing the position of the patient — Patients in the experimental group underwent oropharyngeal aspiration prior to each position change in addition to routine nursing care (Endotracheal aspiration in case of indication and oropharyngeal aspiration in the follow-up; routine and non-routine position changes every 2 hours during the day and 4 hours during the night; oral care).
  Patients in this group underwent oropharyngeal aspiration at least 9 times in 24 hours with a pressure of 100-120 mmHg for 10 seconds prior to routine (2 hours a day, 4 hours a night) and non-routine position changes. After the oropharyngeal aspiration was completed, the patient's position was changed.
  Arms: Experimental group:
Other: Control group: — The patients in the control group received routine nursing care in the unit. (Endotracheal aspiration in case of indication and oropharyngeal aspiration in the follow-up; routine and non-routine position changes every 2 hours during the day and 4 hours during the night; oral care).
  Arms: Control group

SUMMARY:
Ventilator-associated pneumonia (VAP) is one of the healthcare-related infections that is common in critically ill patients, prolongs hospital stay, significantly increases mortality and additional health care costs.

Microaspiration of oropharyngeal secretions the primary pathway in the formation of VAP has led researchers to focus on the detection of applications to prevent microbial colonization. Continuous or intermittent oropharyngeal aspiration, open system aspiration versus closed system aspiration, extensive oral care, oropharyngeal aspiration prior to patient positioning are some of these applications.

When the patient is turned to position, the outbreak accumulated in the oral cavity is more likely to move to the lower respiratory tract. In this study, it is assumed that aspiration of oropharyngeal secretions prior to each position change will reduce the accumulation of oral secretion in the endotracheal tube cuff and reduce aspiration of contaminated secretion and reduce the risk of developing VIP. This randomized controlled experimental study was planned to confirm the validity of this assumption.

This study was a randomized controlled experimental study designed to investigate the effect of oropharyngeal aspiration on decreasing the incidence of ventilator-associated pneumonia in patients receiving mechanical ventilation. The research was conducted between July 2015 and April 2019 in anesthesiology and reanimation intensive care unit. The study was carried out with 20 patients who underwent oropharyngeal aspiration as needed and 20 patients with oropharyngeal aspiration prior to each change of position.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Supported mechanical ventilation by endotracheal tube,
* ≥ 24 hours remaining connected to mechanical ventilator,
* Position can be changed every 2 hours during the day and 4 hours at night,
* Patients whose relatives were approved to participate in the study.

Exclusion Criteria:

* Pneumonia develops prior to mechanical ventilation support or within the first 48 hours following mechanical ventilation support,
* Positive sputum culture was taken before mechanical ventilation support or within the first 48 hours following mechanical ventilation support,
* Patients with diabetes mellitus,
* Patients with contraindications for routine change of position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 20 male and 20 female patients were included in the study.
Enrollment: 40 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Ventilator-Related Pneumonia | Through study completion, about four years]
  Clinical Pulmonary Infection Score (CPIS) was used in the diagnosis of VAP and, VAP was diagnosed in patients whose CPIS was above 6 in the evaluation. Broncho alveolar lavage specimens were cultured for VAP agent/s. Antibiotic susceptibility of microorganisms grown in positive cultures were investigated.

IPD SHARING:
Plan to Share IPD: No